CLINICAL TRIAL: NCT01519661
Title: A Single Arm, Open-label, Multicenter, Phase IV Trial to Assess Long Term Safety of Tobramycin Inhalation Powder (TIP) in Patients With Cystic Fibrosis
Brief Title: Long Term Safety of Tobramycin Inhalation Powder in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTBM100C2401; 2011-002000-32 (EudraCT Number)
Record Dates: First submitted 2012-01-24; First posted 2012-01-27 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Pulmonary Infections; Pseudomonas Aeruginosa in Cystic Fibrosis
Keywords: Tobramycin Inhalation powder; Cystic fibrosis; Lung disease; Anti-bacterial agents
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases

ARMS (1):
- Tobramycin Inhalation Powder (TIP) (Experimental): Eligible patients were assigned to four capsules of TIP at 28mg dosage strength, inhaled b.i.d. in the morning and in the evening via the T-326 inhaler, for 28 days (on treatment), followed by 28 days of no study treatment (off treatment). Each treatment therefore consisted of 112mg tobramycin (4 capsules of 28mg each) with the total daily dose = 224mg tobramycin (112mg b.i.d.). These 56 days represented 1 cycle of therapy.
  Interventions: Drug: TBM100

INTERVENTIONS:
Drug: TBM100 — Tobramycin inhalation powder was assigned as four capsules at 28mg dosage strength. It was inhaled b.i.d in the morning and in the evening via the T-326 Inhaler.

SUMMARY:
This study assessed the long term safety data for the use of tobramycin inhalation powder in patients suffering from cystic fibrosis who have a chronic pulmonary infection with Pseudomonas aeruginosa.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Cystic Fibrosis
* FEV1 at screening must be between 25 and 75 percent of normal predicted values for age, sex and height based on the Knudson equation
* Pseudomonas aeruginosa must be present in a sputum / deep cough throat swab culture or bronchoalveolar lavage within 6 months prior to screening and in the sputum/deep-throat cough swab culture at screening

Exclusion Criteria:

* History of sputum culture or deep cough throat swab culture yielding Burkholderia cenocepacia complex within 2 years prior to screening and /or sputum culture yielding Burkholderia cenocepacia at screening
* Hemoptysis more than 60mL at any time within 30 days prior to study drug administration
* History of hearing loss or chronic tinnitus deemed clinically significant
* Serum creatinine 2mg/dl or more, BUN 40mg/dl or more, or an abnormal urinalysis defined as 2+ or greater proteinuria at screening
* Known local or systemic hypersensitivity to aminoglycosides or inhaled antibiotics
* Patients who are regularly receiving more than 1 class of inhaled anti-pseudomonal antibiotic
* Any use of inhaled or systemic anti-pseudomonal antibiotic within 28 days prior to study drug administration
* Use of loop diuretics within 7 days prior to study drug administration

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (48):
- United States (19):
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Morristown, New Jersey
  - Novartis Investigative Site, Akron, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Tacoma, Washington
  - Novartis Investigative Site, Madison, Wisconsin
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Argentina (4):
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Capital Federal, Buenos Aires
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Paraná, Entre Ríos Province
- Australia (3):
  - Novartis Investigative Site, New Lambton Heights, New South Wales
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Parkville, Victoria
- Canada (3):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Montreal, Quebec
- France (5):
  - Novartis Investigative Site, Giens
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Roscoff
- Germany (2):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
- Novartis Investigative Site, Budapest, Hungary
- Italy (7):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Palermo, Italy
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Roma
- Mexico (2):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia

REFERENCES:
- [Derived] Sommerwerck U, Virella-Lowell I, Angyalosi G, Viegas A, Cao W, Debonnett L. Long-term safety of tobramycin inhalation powder in patients with cystic fibrosis: phase IV (ETOILES) study. Curr Med Res Opin. 2016 Nov;32(11):1789-1795. doi: 10.1080/03007995.2016.1211516. Epub 2016 Sep 9. PMID 27435882

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tobramycin Inhalation Powder (TIP)
Started | 157
Completed | 96
Not Completed | 61
Not completed — Protocol deviation | 6
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 17
Not completed — Lack of Efficacy | 6
Not completed — Adverse Event | 29

BASELINE CHARACTERISTICS:
Arm/Group | Tobramycin Inhalation Powder (TIP)
Number analyzed (Participants) | 157
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.8 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 97
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 57.4 (13.52)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 20.5 (3.35)
FEV1 % predicted [Mean (Standard Deviation); unit: percent] | 50.2 (13.95)
FVC % predicted [Mean (Standard Deviation); unit: percent] | 73.9 (15.88)
FEF25-75 % predicted [Mean (Standard Deviation); unit: percent] | 21.8 (12.75)
Sputum density of P. aeruginosa - sum of all biotypes [Mean (Standard Deviation); unit: log10 Colony Forming Units (CFU)] | 7.6 (1.65)
P. aeruginosa tobramycin minimal inhibitory concentration (MIC) [Number; unit: percentage of participants]
  > 8 ug/mL | 26.1
  <= 8 ug/mL | 73.2
  Missing | 0.6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events, Serious Adverse Events (SAEs) and Deaths
Description: Adverse events were deemed treatment-emergent if the onset date/time was on or after the date and time of first study drug. All adverse events were included after this time during both on and off-treatment periods.
Time Frame: 337 days
Population: Safety set: The safety set included all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Tobramycin Inhalation Powder (TIP)
Number analyzed (Participants) | 157
Percentage of participants
  Adverse events (serious and non-serious) | 85.4
  Serious adverse events | 31.2
  Deaths | 0.0

2. Secondary Outcome: Relative Change From Baseline in Forced Expiratory Volume in One Second (FEV1) Percent Predicted
Description: Spirometry was performed at each visit. FEV1, FVC, and FEF25-75 were recorded at all visits according to American Thoracic Society (ATS) guidelines. FEV1 = the volume of air expired in 1 second. FEV1 % predicted is a normalized value of FEV1 calculated using the Knudsen equation, based upon participant's age, gender and height. FVC (forced vital capacity) = the maximal volume of air exhaled with maximally forced effort from a position of maximal inspiration. FEF25-75 = forced expiratory flow from 25% to 75% of the FVC. Relative change in FEV1 % predicted from baseline to pre-dose day X = ((pre-dose day X FEV1 % predicted - baseline FEV1 % predicted) / baseline FEV1 % predicted) • 100.
Time Frame: Baseline, day 29, day 85, day 141, day 197, day 253, day 309, day 337. All study visits except baseline and day 337 occurred at the end of a 28-day on-treatment period of a cycle. Day 337 was the end of the final 28-day off treatment period.
Population: Participants from the safety set who had FEV1 percent predicted values at both baseline and the post baseline time points were analyzed at each given time point. The safety set included all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tobramycin Inhalation Powder (TIP)
Number analyzed (Participants) | 157
Percent change
  Day 29, Cycle 1 (n=149) | 0.8 (17.17)
  Day 85, Cycle 2 (n=146) | 0.0 (17.09)
  Day 141, Cycle 3 (n=128) | 0.2 (15.13)
  Day 197, Cycle 4 (n=116) | -0.2 (15.36)
  Day 253, Cycle 5 (n=105) | -1.5 (17.19)
  Day 309, Cycle 6 (n=100) | -1.9 (14.55)
  Day 337, Completion (n=93) | -3.5 (16.81)

3. Secondary Outcome: Relative Change From Baseline in FVC Percent Predicted
Description: Spirometry was performed at each visit. FEV1, FVC, and FEF25-75 were recorded at all visits according to American Thoracic Society (ATS) guidelines. FEV1 = the volume of air expired in 1 second. FEV1 % predicted is a normalized value of FEV1 calculated using the Knudsen equation, based upon participant's age, gender and height. FVC (forced vital capacity) = the maximal volume of air exhaled with maximally forced effort from a position of maximal inspiration. FEF25-75 = forced expiratory flow from 25% to 75% of the FVC. Relative change in FVC % predicted from baseline to pre-dose day X = ((pre-dose day X FVC % predicted - baseline FVC % predicted) / baseline FVC % predicted) • 100.
Time Frame: as for outcome 2
Population: Participants from the safety set who had values at both baseline and the given assessment day were included in the analysis for that assessment day. Therefore, the 'n' for each assessment day is different. The safety set included all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tobramycin Inhalation Powder (TIP)
Number analyzed (Participants) | 157
Percent change
  Day 29, Cycle 1 (n=149) | -2.5 (12.95)
  Day 85, Cycle 2 (n=146) | -2.8 (12.81)
  Day 141, Cycle 3 (n=128) | -2.1 (12.25)
  Day 197, Cycle 4 (n=116) | -1.8 (12.64)
  Day 253, Cycle 5 (n=105) | -3.5 (13.11)
  Day 309, Cycle 6 (n=100) | -3.1 (12.17)
  Day 337, Completion (n=93) | -2.8 (13.50)

4. Secondary Outcome: Relative Change From Baseline in FEF Rate Over 25 to 75 Percent of Vital Capacity Predicted
Description: Spirometry was performed at each visit. FEV1, FVC, and FEF25-75 were recored at all visits according to American Thoracic Society (ATS) guidelines. FEV1 = the volume of air expired in 1 second. FEV1 % predicted is a normalized value of FEV1 calculated using the Knudsen equation, based upon participant's age, gender and height. FVC (forced vital capacity) = the maximal volume of air exhaled with maximally forced effort from a position of maximal inspiration. FEF25-75 = forced expiratory flow from 25% to 75% of the FVC. Relative change in FEEF25-75 from baseline to pre-dose day X = ((pre-dose day X FEF25-75 - baseline FEF25-75) / baseline FEF25-75) • 100.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tobramycin Inhalation Powder (TIP)
Number analyzed (Participants) | 157
Percent change
  Day 29, Cycle 1 (n=149) | 10.3 (36.05)
  Day 85, Cycle 2 (n=146) | 9.4 (55.35)
  Day 141, Cycle 3 (n=128) | 5.5 (31.82)
  Day 197, Cycle 4 (n=116) | 6.0 (30.96)
  Day 253, Cycle 5 (n=105) | 2.9 (33.23)
  Day 309, Cycle 6 (n=100) | 4.3 (32.44)
  Day 337, Completion (n=93) | 0.7 (33.78)

5. Secondary Outcome: Change From Baseline in Pseudomonas Aeruginosa Colony Forming Units in Sputum
Description: Sputum was collected in sterile containers and cultured for Pseudomonas aeruginosa (Pa.) (quantitative test) and other typical Cystic Fibrosis respiratory pathogens. The Pa. biotypes measured were mucoid, dry and small colony variant. Results are presented for the sum of all biotypes of Pa, with data transformed using a base 10 logarithm.
Time Frame: Baseline, day 1, day 29, day 85, day 141, day 197, day 253, day 309, day 337
Population: Participants from the safety set who had Pa sputum density values at both baseline and the given time point were included in the analysis. The safety set included all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: log10 Colony Forming Unit (CFU)
Arm/Group | Tobramycin Inhalation Powder (TIP)
Number analyzed (Participants) | 157
log10 Colony Forming Unit (CFU)
  Sum of all biotypes, Day 29, Cycle 1 (n=141) | -1.6 (2.28)
  Sum of all biotypes, Day 85, Cycle 2 (n=135) | -1.1 (1.80)
  Sum of all biotypes, Day 141, Cycle 3 (n=119) | -1.2 (1.98)
  Sum of all biotypes, Day 197, Cycle 4(n=107) | -1.1 (2.11)
  Sum of all biotypes. Day 253, Cycle 5 (n=98) | -1.3 (2.23)
  Sum of all biotypes, Day 309, Cycle 6 (n=89) | -1.2 (2.09)
  Sum of all biotypes, Day 337, Completion (n=85) | -0.4 (2.08)

6. Secondary Outcome: Tobramycin MIC 50 and MIC 90 Values Over All Isolates for the Sum of All Biotypes (Mucoid, Dry and Small Colony Variant) of Pseudomonas Aeruginosa
Description: Tobramycin MIC 50 and MIC 90 values were defined as the lowest concentration of tobramycin required to inhibit 50% and 90%, respectively, of the P. aeruginosa strains tested.
Time Frame: Baseline, day 29, day 85, day 141, day 197, day 253, day 309, day 337
Population: Participants from the safety set who had data at each time point/cycle were analyzed at each time point. The safety set included all participants who received at least one dose of study drug.
Measure: Number; unit: ug/mL
Groups:
- Tobramycin Inhalation Powder (TIP): Eligible patients were assigned to four capsules of TIP at 28mg dosage strength, inhaled b.i.d. in the morning and in the evening via the T-326 inhaler, for 28 days (on treatment), followed by 28 days of no study treatment (off treatment). Each treatment therefore consisted of 112mg tobramycin (4 capsules of 28mg each) with the total daily dose = 224mg tobramycin (112mg b.i.d.). These 56 days represented 1 cycle of therapy. Total number of isolates at each cycle/day: baseline = 279; cycle 1, day 29 = 252; cycle 2, day 85 = 238; cycle 3, day 141 = 210; cycle 4, day 197 = 184; cycle 5, day 253 = 178; cycle 6, day 309 = 164; and completion, day 337 = 158
Arm/Group | Tobramycin Inhalation Powder (TIP)
Number analyzed (Participants) | 157
ug/mL
  Baseline - MIC 50 (n=156) | 2
  Cycle 1, day 29 - MIC 50 (n=144) | 2
  Cycle 2, day 85 - MIC 50 (n=137) | 2
  Cycle 3, day 141 - MIC 50 (n=124) | 2
  Cycle 4, day 197 - MIC 50 (n=108) | 2
  Cycle 5, day 253 - MIC 50 (n=98) | 2
  Cycle 6, day 309 - MIC 50 (n=90) | 4
  Completion, day 337 - MIC 50 (n=89) | 2
  Baseline - MIC 90 (n=156) | 128
  Cycle 1, day 29 - MIC 90 (n=144) | 256
  Cycle 2, day 85 - MIC 90 (n=137) | 256
  Cycle 3, day 141 - MIC 90 (n=124) | 256
  Cycle 4, day 197 - MIC 90 (n=108) | 128
  Cycle 5, day 253 - MIC 90 (n=98) | 256
  Cycle 6, day 309 - MIC 90 (n=90) | 256
  Completion, day 337 - MIC 90 (n=89) | 512

7. Secondary Outcome: Percentage of Participants Hospitalized Due to Serious Respiratory-related Adverse Events
Time Frame: Day 337
Population: Safety set: The safety set included all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Tobramycin Inhalation Powder (TIP)
Number analyzed (Participants) | 157
Percentage of participants | 26.8

8. Secondary Outcome: Number of Hospitalization Days Due to Serious Respiratory-related Adverse Events
Description: The total number of hospitalization days due to serious respiratory-related adverse events was analyzed.
Time Frame: Day 337
Population: Safety set: The safety set included all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Tobramycin Inhalation Powder (TIP)
Number analyzed (Participants) | 157
Days | 18.1 (17.14)

9. Secondary Outcome: Time to First Hospitalization Due to Serious Respiratory-related Adverse Events
Description: The day of first hospitalization due to serious respiratory-related adverse events was analyzed.
Time Frame: Day 337
Population: Safety set The safety set included all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tobramycin Inhalation Powder (TIP)
Number analyzed (Participants) | 157
Days | NA [NA to NA] — The median was not estimable due to an insufficient number of events.

10. Secondary Outcome: Percentage of Participants Who Used New Anti-pseudomonal Antibiotics
Time Frame: Day 337
Population: Safety set: The safety set included all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Tobramycin Inhalation Powder (TIP)
Number analyzed (Participants) | 157
Percentage of participants | 65.6

11. Secondary Outcome: Number of Days of New Anti-pseudomonal Antibiotic Use
Description: The total number of days of new anti-pseudomonal antibiotic use was analyzed.
Time Frame: Day 337
Population: Safety set: The safety set included all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Tobramycin Inhalation Powder (TIP)
Number analyzed (Participants) | 157
Days | 33.1 (25.17)

12. Secondary Outcome: Time to Use of New Anti-pseudomonal Antibiotic
Description: Time to first use of new anti-pseudomonal antibiotic was analyzed.
Time Frame: Day 337
Population: Safety set The safety set included all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tobramycin Inhalation Powder (TIP)
Number analyzed (Participants) | 157
Days | 136 [97 to 170]

ADVERSE EVENTS:
Arm/Group | Tobramycin Inhalation Powder (TIP)
Serious Adverse Events (participants affected / at risk) | 49/157
Other Adverse Events (participants affected / at risk) | 121/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tobramycin Inhalation Powder (TIP) (N=157)
Supraventricular tachycardia (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Deafness unilateral (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Bronchopneumonia (Infections and infestations) | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 39
Influenza (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 3
Rib fracture (Injury, poisoning and procedural complications) | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tobramycin Inhalation Powder (TIP) (N=157)
Abdominal pain (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 7
Chest discomfort (General disorders) | 9
Fatigue (General disorders) | 9
Pyrexia (General disorders) | 12
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 66
Nasopharyngitis (Infections and infestations) | 20
Pharyngitis (Infections and infestations) | 5
Rhinitis (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 15
Forced expiratory volume decreased (Investigations) | 8
Headache (Nervous system disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 37
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 33
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 5
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 16
Wheezing (Respiratory, thoracic and mediastinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.